CLINICAL TRIAL: NCT00747097
Title: Gemcitabine and Cetuximab in Patients With Advanced or Metastatic Biliary Tract Cancer: A Multicenter Phase II Study
Acronym: ECHO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Ivan Borbath, MD, BGDO
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 62202-788
Record Dates: First submitted 2008-09-03; First posted 2008-09-04 (Estimated); Last update posted 2011-02-10 (Estimated); Status verified 2011-02

CONDITIONS: Time to Progression
MeSH Terms: interventions — Gemcitabine; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): gemcitabine+cetuximab
  Interventions: Drug: gemcitabine + cetuximab

INTERVENTIONS:
Drug: gemcitabine + cetuximab — gemcitabine 1g/m² 3weeks/4 cetuximab 400 mg/m² the first week, then 250 mg/m², every week Every cycle is 8 weeks treatment

SUMMARY:
The purpose of this phase II study is to assess the efficacy of combined chemotherapy using gemcitabine and cetuximab for advanced cholangiocarcinoma, excluding gallbladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically proven locally advanced or metastatic unresectable adenocarcinoma of the biliary tract
* signed written informed consent
* age > 18
* WHO PS 0 or 1 at study entry
* measurable (diameter ³ 1 cm) / evaluable disease, according to RECIST criteria
* adequate renal (serum creatinin<1.5x upper reference range), liver (total bilirubin<2x upper reference range) and hematopoietic functions (PMN>1,5x109/L, platelets>100x109/L)
* life expectancy of at least 12 weeks
* effective contraception throughout the study for both male and female patients if the risk of conception exists

Exclusion Criteria:

* uncontrolled concurrent CNS, cardiac, infectious diseases
* previous exposure to epidermal growth factor targeting therapy
* known hypersensitivity to any components of study treatments
* previous chemotherapy for this cancer
* previous malignancy in the last past 5 years except basal cell cancer of the skin or preinvasive cancer of the cervix
* pregnancy or breast feeding
* medical or psychological conditions that would not permit the patient to complete the study or sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 6 months

SECONDARY OUTCOMES:
overall survival, objective response, safety | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques Universitaires St.-Luc, Brussels, Belgium

REFERENCES:
- [Derived] Borbath I, Ceratti A, Verslype C, Demols A, Delaunoit T, Laurent S, Deleporte A, Vergauwe P, Van Maanen A, Sempoux C, Van Cutsem E, Van Laethem JL; Belgian Group of Digestive Oncology. Combination of gemcitabine and cetuximab in patients with advanced cholangiocarcinoma: a phase II study of the Belgian Group of Digestive Oncology. Ann Oncol. 2013 Nov;24(11):2824-9. doi: 10.1093/annonc/mdt337. Epub 2013 Aug 23. PMID 23975665